CLINICAL TRIAL: NCT03464032
Title: A Multicenter Open-Label Single-Arm Multi-Cohort Phase I Study of Pharmacokinetics, Safety, and Immunogenicity of BCD-135 (JSC BIOCAD, Russia) in Patients With Advanced Solid Tumors
Brief Title: A Study of BCD-135 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCD-135-1
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Melanoma; NSCLC; Renal Cell Carcinoma; Bladder Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD-135 (Experimental): Dose-escalation Arm (0.4, 1, 3, 10, 20 mg/kg)
  Interventions: Drug: BCD-135

INTERVENTIONS:
Drug: BCD-135 — Monoclonal anti-PD-L1 antibody

SUMMARY:
A Multicenter Open-Label Single-Arm Multi-Cohort Phase I Study of Pharmacokinetics, Safety, and Immunogenicity of BCD-135 (JSC BIOCAD, Russia) in Patients with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides a written informed consent and is able to follow the requirements of the Protocol;
2. Age ≥ 18 years
3. Histologically confirmed cancer (well-documented test results; preferably, block specimens available):

   * Unresectable (stage III/IV) or metastatic (stage IV) melanoma (the drug will be used as the first or subsequent therapy lines);
   * Locally advanced or metastatic EGFR/ALK wt NSCLC (squamous cell carcinoma/adenocarcinoma), progressive after the first-line therapy with platinum-based CT or EGFR/ALK wt NSCLC progressive after the first-line therapy with EGFR/ALK inhibitors (the drug will be used as a second therapy line);
   * Metastatic clear cell renal carcinoma, progressive after at least the first-line therapy (the drug will be used as a second or third therapy lines);
   * Locally advanced or metastatic bladder cancer progressive on/after therapy with platinum-based CT (the drug will be used as a second therapy line);
4. ECOG score of 0 to 1;
5. Presence of blocks for histological examination and/or patient's agreement to conduct a biopsy of an accessible lesions to obtain a histological material for examination of PD-L1 status
6. Measurable disease (at least one lesion) according to RECISTv.1.1;
7. Resolved toxicity events from the previous therapy or adverse consequences of surgical interventions to ≤ grade 1 CTCAE v. 4.03, except for chronic/irreversible adverse events not affecting the safety of the study therapy (e.g. alopecia);
8. No severe pathology of organs or systems;
9. Life expectancy of at least 12 weeks from the screening;
10. Patients of childbearing potential enrolled in the study must agree to use reliable contraception methods throughout the study period, beginning 2 weeks before the inclusion in the study and up to 8 weeks after the last dose of BCD-100.

Exclusion Criteria:

1. Severe concomitant illnesses or life-threatening consequences (including pleural/pericardial/peritoneal effusion that requires medical intervention, pulmonary lymphangitis, or involvement of >50% renal parenchyma);
2. Brain metastases, progressive or associated with clinical symptoms (e.g. cerebral edema or spinal cord compression). Exclusions: metastases that do not progress and do not require steroids and/or anticonvulsants within at least 4 weeks before randomization;
3. Severe cardiovascular disorders within 6 months before screening;
4. Autoimmune diseases;
5. Conditions requiring steroids or any other immunosuppressants;
6. Blood disorders: ANC ≤1,500/mm3; platelets ≤100,000/mm3; or Hb ≤90 g/L;
7. Renal function impairment: creatinine ≥1.5 × ULN;
8. Hepatic function impairment: bilirubin ≥1.5 × ULN; AST and ALT ≥2.5 × ULN (5 × ULN for patients with liver metastases), AlkPh ≥ 5 × ULN;
9. LDH level >2 ULN;
10. Prior anticancer treatment within 28 days before starting the study drug (surgery, radiation therapy, targeted therapy, immunotherapy, vaccine treatment or chemotherapy);
11. More than

    * 2 therapy lines of unresectable/metastatic melanoma,
    * 1 therapy line of metastatic NSCLC,
    * 2 therapy lines of metastatic RCC;
    * 1 therapy line of metastatic BC;
12. Prior treatment with anti-PD1/PDL1 agents or CTLA4 inhibitors;
13. Concurrent malignancy except for radically resected cervical carcinoma in situ or radically resected basal cell/squamous cell carcinoma;
14. Conditions limiting patient's ability to follow the Protocol requirements (dementia, neurological or psychiatric disorders, drug or alcohol abuse, etc.);
15. Simultaneous participation in any other clinical trial; participation in other clinical trials within 28 days before inclusion in the present study; previous participation in the present study.
16. Acute infections or active chronic infections;
17. Documented HIV infection;
18. Positive screening results for Hbs-antigen, hepatitis B core antibodies (anti-HBc Ab) and/or hepatitis C antibodies;
19. Positive results of microprecipitation reaction together with positive TPHA assay results at the screening;
20. Body weight > 100 kg.
21. Intravenous administration of the drug is impossible;
22. Intravenous administration of contrast agents is impossible;
23. Hypersensitivity to any component of BCD-100.
24. Known history of hypersensitivity to monoclonal antibodies;
25. Pregnancy or breastfeeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
DCR | 85 days
  Disease control rate (CR+PR+SD). Pilot efficacy assessment is not the primary objective of this study and will be conducted by surrogate endpoints describing the direct antitumor effect of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Odintsova, MD, Principal Investigator — LLC BioEk
Locations (1):
- LLC BioEk, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided